CLINICAL TRIAL: NCT01656005
Title: Evaluation of Effects of Chronic Dose Exposure to Cardioselective and Non-cardioselective Beta Blockers on Measures of Cardiopulmonary Function in Moderate to Severe COPD.
Brief Title: Beta Blocker Therapy in Moderate to Severe COPD
Acronym: ANDA2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Tenovus Scotland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANDA2; 2011-006008-11 (EudraCT Number)
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Beta blockers; Cardioselective; Non-cardioselective; Impulse oscillometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Carvedilol; Bisoprolol; Beclomethasone; Formoterol Fumarate; Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol (Experimental): Beclometasone/Formoterol Beclometasone Tiotropium
  Interventions: Drug: Carvedilol; Drug: Beclometasone/formoterol; Drug: Tiotropium; Drug: Beclometasone
- Bisoprolol (Active Comparator): Beclometasone/Formoterol Beclometasone Tiotropium
  Interventions: Drug: Bisoprolol; Drug: Beclometasone/formoterol; Drug: Tiotropium; Drug: Beclometasone

INTERVENTIONS:
Drug: Carvedilol — Dose titration: 3.125mg bid for 1 week, 6.25mg bid for 1 week, 12.5mg bid for 4 weeks.
  Arms: Carvedilol
Drug: Bisoprolol — Dose titration: 1.25mg od for 1 week, 2.5mg od for 1 week, 5mg for 4 weeks.
  Arms: Bisoprolol
Drug: Beclometasone/formoterol — 2 puffs bid for first 5 weeks in each treatment arm
  Other Names: Fostair 100/6
Drug: Tiotropium — 1 puff daily for first 4 weeks of each treatment arm
  Other Names: Spiriva 18mcg
Drug: Beclometasone — 2 puffs bid for final week (week 6) of each treatment arm
  Other Names: Clenil 200

SUMMARY:
Beta blockers are a type of medication mainly used for heart disease. They are commonly used to treat 'angina' and to prevent heart attacks. Patients with COPD are more likely to suffer from heart disease and so already benefit from this treatment for this reason. In addition to this, new research suggests that there may be further benefit of using beta blockers for COPD, even without also having heart disease.

The reason why beta blockers are not widely used in COPD at present is because of their potential to make symptoms of COPD worse by causing the airways to narrow. Beta blockers are the opposite type of medication to 'beta-agonists' such as salbutamol which you may be taking for symptoms of breathlessness or wheezing. Nevertheless beta blockers are still used in COPD where the benefits (for example heart disease) outweigh any risks.

Current COPD treatment includes inhaled steroids and long acting beta agonists, often given in a combination inhaler (e.g. Seretide or Symbicort) to treat both airway inflammation and airway narrowing, leading to improvement in symptoms. Another drug commonly used is Tiotropium (Spiriva) which is another type of long acting inhaler medication to help with widening the airways.

In this study, we wish to find out if two different types of beta blocker cause different effects on the airways in COPD patients. One type of beta blocker is more 'selective' in acting mainly on the heart, with the other type having more general or 'non-selective' effects on both the heart and lungs. By doing this we will also be able to look at how the beta blockers work alongside the 'usual' inhaler treatment described above.

DETAILED DESCRIPTION:
Screening Visit A member of the research team will discuss the Patient Information Sheet with the participant, answer any questions posed and written informed consent will be obtained.

Prior to screen participants will be asked to withhold tiotropium for 48 hours ipratropium bromide for 12 hours and salbutamol for 6 hours.

A general physical examination will be carried out by a qualified medical practitioner.

A pregnancy test from a urine sample will be performed for all female participants with advice issued to both male and female participants to use contraception throughout the duration of the study.

The following will be measured:

Spirometry with sequential reversibility to 400μg salbutamol then 80 μg ipratropium bromide according to American Thoracic Society guidelines Resting Electrocardiogram Whole body plethysmography (where possible) Impulse Oscillometry

Oxygen saturations breathing room air after 5 mins rest Heart rate and blood pressure. 6 Minute Walk Test (if physically able)

Inhaler technique will be assessed and confirmed adequate.

Full blood count, renal function, electrolytes, liver enzymes and random blood glucose will be measured.

Participants will be checked against all inclusion and exclusion criteria. Those found to be eligible will proceed to the run-in period.

Run-in period Participants who are taking inhaled corticosteroids, combination inhalers, Long acting bata agonists or long-acting anti-muscarinics will have these discontinued.

All participants entering the run-in period will be commenced on Fostair (Beclometasone/Formoterol) 100/6, 2 puffs twice daily via spacer device for approximately 2 weeks.

Participants will be given a PiKO monitor to record domiciliary Forced expiratory volume1 and Forced expiratory Volume6 twice daily (approximately 12 hours apart) in a diary supplied by the department as well as domiciliary oxygen saturation and Heart Rate monitor to be recorded twice daily. They will also complete a daily diary of reliever use and symptoms. These will all be performed from the beginning of the run-in period to the end of the study.

At the end of run-in, participants will be again checked against all inclusion and exclusion criteria and the hief Investigator or medical investigator for the study will sign the declaration on the Case Report Form, to confirm the subject's suitability to receive the study drug according to study protocol. Those eligible will proceed to study visit 1. Those who do not fulfil the study criteria will be returned to their pre-study medication and their GP informed of any medically relevant data.

Study Visit 1 (Baseline 1) Participants will attend the department on the morning of their study visit.

Participants will be asked to withhold their ipratropium for 12 hours and salbutamol for 6 hours prior to visit.

Diaries of symptoms, reliever use and domiciliary FEV1 will be reviewed.

Baseline measurements to be recorded are:

IOS Slow Vital Capacity Spirometry Resting ECG Resting O2 sats HR and BP St George's Respiratory Questionnaire 6MWT (where physically possible and only if performed at screen) Echocardiogram (where technically possible) Serum (after at least 30mins supine posture): Aldosterone, Angiotensin II, BDNF, BNP, Potassium

Provided average HR>60bpm and average systolic BP>110mmHg the participant will be randomised to 1 of 2 beta-blocker treatments comprising:

1. Carvedilol: 1 week of 3.125mg bid, 1 week of 6.25mg bid, 4 weeks of 12.5mg bid or
2. Bisoprolol: 1 week of 1.25mg od, 1 week of 2.5mg od, 4 weeks of 5mg od

Participants will be given their first 4 weeks of randomised IMP for the treatment period at this study visit.

When titrating their beta-blocker at home, should the participant start to experience side-effects related to beta-blocker therapy or they find that their HR is dropping below 55bpm they will be informed to phone the department working hours) or the emergency mobile number (out of hours).

Participants will be allowed to complete each treatment arm on their maximum tolerated dose of beta-blocker, should this be less than the maximum prescribed dose.

Participants in both treatment arms will continue taking Fostair 100/6, 2 puffs bid via spacer device for the first 5 weeks of each treatment period. For the final (6th) week of each treatment period they will receive inhaled beclometasone dipropionate (as Clenil) 200μg, 2 puffs bid via spacer device, instead of Fostair.

Participants in both treatment arms will be given Tiotropium 18μg (via handihaler) od for the first 4 weeks of each treatment period. Tiotropium will then be discontinued for the final 2 weeks of each treatment period.

Participants will be given a salbutamol inhaler to use as initial reliever therapy along with an ipratropium inhaler second line on a PRN basis.

The IMPs will be issued to the participant by a member of the research team delegated the task. The allocation will be checked and countersigned by a second delegated member of staff.

Inhaler technique for the different devices will be checked.

A participant instruction and appointment leaflet will be issued and discussed fully with the participant and any questions answered. It will detail:

Emergency contact numbers Instructions on how to take heart rate and O2 sats measurements How to perform domiciliary FEV1 and FEV6 How to write in the diary Potential side effects of study drugs Recording of AEs and concomitant medication use Withholding times for relievers Titration/Discontinuation times for IMPs

Reminders to return medication and bottles at each visit

Study visit 2

Measurements to be recorded at this visit are:

IOS Slow VC Spirometry Resting O2 sats HR and BP (as previously described in 3.5.5) Resting ECG 6MWT (where physically possible and only if performed previously in study) SGRQ

Participants will be given their final 2 weeks of randomised IMP (at their maximum tolerated dose) for that treatment period.

Participants will discontinue their tiotropium for the remaining 2 weeks of the treatment period at this study visit.

Study visit 3

. As for study visit 2 with the addition of Serum BDNF, Potassium

Participants will discontinue their Fostair inhaler at this study visit and be given Clenil (beclometasone) 200ug, 2 puffs bid to take instead for the final week of the treatment period.

Study visit 4 As before plus, Echocardiogram (where technically possible) Serum (after at least 30mins supine posture): Aldosterone, Angiotensin II, BDNF, BNP, Potassium

Participants will finish treatment period 1 at this point and enter a 2 week period of washout (of beta-blocker) prior to crossing over to the other treatment arm.

Participants will discontinue their Clenil and beta-blocker and return to taking Fostair 100/6, 2 puffs bid for the 2 week washout period.

Study Visit 5 (Baseline 2)

Measurements to be recorded are:

IOS Slow VC Spirometry Resting ECG Resting O2 sats HR and BP (as previously described in 3.5.5) SGRQ 6MWT (where physically possible and only if performed at screen) Serum (after at least 30mins supine posture): Aldosterone, Angiotensin II, BDNF, BNP, Potassium

Provided average HR>60bpm and average systolic BP>110mmHg the participant will be crossed over to the beta-blocker treatment that they have not yet received (based on original randomisation) comprising:

1. Carvedilol: 1 week of 3.125mg bid, 1 week of 6.25mg bid, 4 weeks of 12.5mg bid
2. Bisoprolol: 1 week of 1.25mg od, 1 week of 2.5mg od, 4 weeks of 5mg od Measurements will be repeated as per Study Visit 1.

Study Visits 6 & 7 Visit 6 will be the same as visit 2 Visit 7 will be the same as visit 3 Study Visit 8

Measurements to be recorded are:

IOS Slow VC Spirometry Resting ECG Resting O2 sats HR and BP (as previously described in 3.5.5) SGRQ 6MWT (where physically possible and only if performed at screen) Echocardiogram (where technically possible) Serum (after at least 30mins supine posture): Aldosterone, Angiotensin II, BDNF, BNP, Potassium

Participants will finish treatment period 2, and, therefore, the study at this point. They will be returned to their usual prescribed medication.

End of Study Period. The study will be complete when the last enrolled participant completes the last visit

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe COPD (GOLD stage 2 and 3)
* FEV1 30-80% predicted
* No exacerbation in previous 3 months
* Smoking history ≥ 10 pack years
* Oxygen saturations≥ 92% on room air at rest
* ECG demonstrating sinus rhythm

Exclusion Criteria:

* Use of domiciliary oxygen
* History of other primary obstructive lung disease including asthma or bronchiectasis
* History of unstable angina, uncontrolled hypertension or heart failure NYHA class 3-4
* Overt clinical signs of right heart failure
* Average resting systolic BP<110mmHg
* Average resting HR<60bpm
* Pregnancy or lactation
* Known or suspected sensitivity to/intolerance of investigational medicinal product
* Inability to comply with compulsory aspects of protocol
* Any degree of heart block
* Concomitant prescription of beta-blockers, rate-limiting calcium channel blockers, digoxin or amiodarone
* Any clinically significant medical condition that may endanger the health or safety of the participant, or jeopardise the protocol
* Participation in another trial within the previous 30 days

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in airway resistance at 5HZ (R5) using impulse oscillometry from baseline. | 4, 5 and 6 weeks of each treatment period

SECONDARY OUTCOMES:
Change in remaining impulse oscillometry measurements from baseline | 4, 5 and 6 weeks of each treatment period
  Resistance at 20Hz (R20); Reactance at 5Hz (X5); Area under reactance curve (Ax); Resonant frequency (Fres).
Change in spirometry measurements from baseline | 4, 5 and 6 weeks of each treatment period
  Forced expiratory volume in 1 sec (FEV1); Forced vital capacity (FVC); Slow vital capacity; Forced expiratory flow between 25-75% of FVC (FEF25-75)
Change in echocardiogram parameters from baseline | At 6 weeks of each treatment period
  Left ventricular function, right ventricular function, pulmonary pressure, pulmonary acceleration time.
Change in vital signs from baseline | 4, 5, and 6 weeks in each treatment period
  Resting oxygen saturations, heart rate, office blood pressure,
Change in six minute walk test distance from baseline | 4, 5 and 6 weeks of each treatment periods.
Change in St George's Respiratory Questionnaire score from baseline | 4, 5 and 6 weeks in each treatment arm

OTHER OUTCOMES:
Daily domiciliary measurements - trends over course of study | Twice daily measurements
  Forced expiatory volume in 1 sec (FEV1); symptom diary; reliever use diary (number of puffs); oxygen saturations; heart rate.
Change in serum B-type natriuretic peptide (BNP) from baseline | 6 weeks in each treatment period
Change in serum aldosterone levels from baseline | 6 weeks in each treatment period
Change in serum angiotensin II levels from baseline | 6 weeks in both treatment arms
Change in serum brain-derived neurotrophic factor (BDNF) from baseline | Weeks 5 and 6 in both treatment periods
Change in serum potassium levels from baseline | Weeks 5 and 6 of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: William J Anderson, MBChB, Principal Investigator — University of Dundee; Brian J Lipworth, MD, Study Director — University of Dundee
Locations (1):
- Asthma and Allergy Research Group, Ninewells Hospital and Medical School, University of Dundee, Dundee, United Kingdom

REFERENCES:
- [Result] Jabbal S, Anderson W, Short P, Morrison A, Manoharan A, Lipworth BJ. Cardiopulmonary interactions with beta-blockers and inhaled therapy in COPD. QJM. 2017 Dec 1;110(12):785-792. doi: 10.1093/qjmed/hcx155. PMID 29025008